CLINICAL TRIAL: NCT00291668
Title: A Phase II, Multi-center, Double-blind, Placebo-controlled, Parallel-group, Dose-response Study to Assess the Safety and Efficacy of CDP870/Certolizumab Pegol, Dosed Subcutaneously in Patients With Active Crohn's Disease
Brief Title: Clinical Study of CDP870/Certolizumab Pegol in Patients With Active Crohn's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C87037; 2014-004399-42 (EudraCT Number)
Record Dates: First submitted 2006-02-10; First posted 2006-02-14 (Estimated); Results first posted 2020-08-03 (Actual); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease; CDP870; Certolizumab pegol
MeSH Terms: conditions — Crohn Disease | interventions — Certolizumab Pegol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Certolizumab pegol 200 mg (Experimental): Subjects received one subcutaneous (sc) injection of 200 mg CZP and one injection of Placebo to maintain the study blind on Weeks 0 (first dose), 2 and 4.
  Interventions: Biological: Certolizumab Pegol; Other: Placebo
- Certolizumab pegol 400 mg (Experimental): Subjects received two subcutaneous (sc) injections of 200 mg CZP on Weeks 0 (first dose), 2 and 4.
  Interventions: Biological: Certolizumab Pegol
- Placebo (Placebo Comparator): Subjects received two subcutaneous (sc) injections of Placebo on Weeks 0 (first dose), 2 and 4.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Certolizumab Pegol — * Active Substance: Certolizumab Pegol
  * Pharmaceutical Form: Solution for injection in pre-filled syringe
  * Concentration: 200 mg/mL
  * Route of Administration: Subcutaneous use
  Other Names: CDP870
  Arms: Certolizumab pegol 200 mg; Certolizumab pegol 400 mg
Other: Placebo — * Active Substance: isotonic sodium chloride solution
  * Pharmaceutical Form: Solution for injection
  * Concentration: 1 mL
  * Route of Administration: Subcutaneous use
  Arms: Certolizumab pegol 200 mg; Placebo

SUMMARY:
This is a multi-centre, randomized, double-blind, dose response clinical study of CDP870 in patients with Crohn's disease.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria:

* Patients who are diagnosed with Crohn's disease (according to the Crohn's disease diagnostic criteria developed by the research group on intractable inflammatory bowel disorders [Shimoyama group, January 25, 2002]) at least 24 weeks before the starting date of the observation period
* Patients with Crohn's Disease Activity Index (CDAI) score ranging from 220 to 450 inclusive during the observation period
* C-reactive protein (CRP) of 1 mg/dL or higher in the laboratory test performed at the start of the observation period

Exclusion Criteria:

* Stoma patient
* Patients with a history of severe hypersensitivity or anphylactic reaction to anti-TNF alpha antibody
* Patients who participated in a clinical study with CDP870
* Pregnant or lactating patients, patients of childbearing potential, or patients who will attempt pregnancy during the study period
* Patients who are judged inappropriate for enrollment by the principal investigator or subinvestigators

Exclusion Criteria:

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2006-03-02 (Actual); Primary Completion 2007-11-08 (Actual); Study Completion 2007-11-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (22):
- Japan (22):
  - Aichi-Gun, Aichi-ken
  - Nagoya, Aichi-ken
  - Toyoake, Aichi-ken
  - Toyohashi, Aichi-ken
  - Kashiwa, Chiba
  - Sakura, Chiba
  - Chikusino, Fukuoka
  - Asahikawa, Hokkaido
  - Sapporo, Hokkaido
  - Nishinomiya, Hyōgo
  - Yokohama, Kanagawa
  - Miyazaki-gun, Miyazaki
  - Kurashiki, Okayama-ken
  - Tyuto-gun, Okinawa
  - Suita, Osaka
  - Ōtsu, Shiga
  - Shinjyuku, Tokyo
  - Fukuoka
  - Kagoshima
  - Nagasaki
  - Niigata
  - Osaka

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study started to enroll subjects in March 2006 and conluded in November 2007.
Pre-assignment Details: Participant Flow refers to the Safety Set, including all randomized subjects who received at least one dose of study medication (Placebo or Certolizumab Pegol).
Period: Overall Study
Arm/Group | Placebo | Certolizumab Pegol 200 mg | Certolizumab Pegol 400 mg
Started | 32 | 30 | 32
Completed | 28 | 29 | 31
Not Completed | 4 | 1 | 1
Not completed — Lack of Efficacy | 1 | 0 | 0
Not completed — SAE, non-fatal | 1 | 1 | 1
Not completed — AE, non-serious non-fatal | 1 | 0 | 0
Not completed — SAE, non-fatal+AE, non-serious non-fatal | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Safety Population, including all randomized subjects who received at least one dose of study medication (Placebo or Certolizumab Pegol).
Arm/Group | Placebo | Certolizumab Pegol 200 mg | Certolizumab Pegol 400 mg | Total Title
Number analyzed (Participants) | 32 | 30 | 32 | 94
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 2 | 2 | 6
  Between 18 and 65 years | 30 | 28 | 30 | 88
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.6 (8.16) | 32.7 (9.34) | 31.4 (8.27) | 31.5 (8.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 7 | 21
  Male | 26 | 22 | 25 | 73

OUTCOME MEASURES:

1. Primary Outcome: Crohn's Disease Activity Index (CDAI) Response (Clinical Response or Remission) at Week 6
Description: CDAI Response is presented as the percentage of subjects with clinical response at Week 6 or remission at Week 6. Clinical response is defined as at least a 100-point decrease from the Week 0 CDAI score, where change = (CDAI score at Week 6) - (CDAI score at Week 0). Remission is defined as a CDAI of <= 150 at Week 6.
Time Frame: Baseline, Week 6
Population: Full Analysis Set defined as subjects randomized and allocated to study medication, excluding the following subjects determined by data review prior to unblinding:
  Subjects
  * with Good Clinical Practice (GCP) violations
  * who were not diagnosed (definitely) with CD
  * who received no dose of study medication
  * with no data after randomization
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Groups:
- Full Analysis Set (Placebo Treated Subjects); Full Analysis Set (CZP 200 mg Treated Subjects); Full Analysis Set (CZP 400 mg Treated Subjects): The Full Analysis Set was defined as the subjects who were randomized and allocated to study medication, but excluded the following subjects as determined by data review prior to unblinding:
  * Subjects with Good Clinical Practice (GCP) violations
  * Subjects who were not diagnosed (definitely) with Crohn's Disease
  * Subjects who received no dose of study medication
  * Subjects with no data after randomization
Arm/Group | Full Analysis Set (Placebo Treated Subjects) | Full Analysis Set (CZP 200 mg Treated Subjects) | Full Analysis Set (CZP 400 mg Treated Subjects)
Number analyzed (Participants) | 32 | 30 | 31
percentage of subjects | 25.0 [10.0 to 40.0] | 43.3 [25.6 to 61.1] | 48.4 [30.8 to 66.0]

2. Secondary Outcome: Crohn's Disease Activity Index (CDAI) Score at Week 2
Description: The Crohn's Disease Activity Index (CDAI) is used to quantify the symptoms of subjects with Crohn's Disease. The CDAI score can range from 0-600 (600 indicating the worst disease). It is the sum of 8 subscores, only the summary score is used here. A CDAI score of 150 or less is considered as remission and a score above 450 indicates extremely severe disease. A decrease in CDAI over time indicates improvement in disease activity.
Time Frame: Week 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Full Analysis Set (Placebo Treated Subjects) | Full Analysis Set (CZP 200 mg Treated Subjects) | Full Analysis Set (CZP 400 mg Treated Subjects)
Number analyzed (Participants) | 29 | 29 | 31
units on a scale | 255.9 (68.02) | 214.2 (83.51) | 224.9 (85.05)

3. Secondary Outcome: Crohn's Disease Activity Index (CDAI) Score at Week 4
Description: as for outcome 2
Time Frame: Week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Full Analysis Set (Placebo Treated Subjects) | Full Analysis Set (CZP 200 mg Treated Subjects) | Full Analysis Set (CZP 400 mg Treated Subjects)
Number analyzed (Participants) | 28 | 27 | 30
units on a scale | 243.1 (68.57) | 199.7 (91.25) | 204.6 (75.10)

4. Secondary Outcome: Crohn's Disease Activity Index (CDAI) Score at Week 6
Description: as for outcome 2
Time Frame: Week 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Full Analysis Set (Placebo Treated Subjects) | Full Analysis Set (CZP 200 mg Treated Subjects) | Full Analysis Set (CZP 400 mg Treated Subjects)
Number analyzed (Participants) | 28 | 27 | 30
units on a scale | 232.4 (89.28) | 211.0 (99.91) | 198.1 (87.88)

5. Secondary Outcome: Percentage of Subjects Who Achieve CDAI Response at Week 2
Description: CDAI Response at Week 2 is defined as clinical response at Week 2 or remission at Week 2. Clinical response is defined as at least a 100-point decrease from the Week 0 CDAI score, where change = (CDAI score at Week 2) - (CDAI score at Week 0). Remission is defined as a CDAI score of <= 150 points.
Time Frame: Baseline, Week 2
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Full Analysis Set (Placebo Treated Subjects) | Full Analysis Set (CZP 200 mg Treated Subjects) | Full Analysis Set (CZP 400 mg Treated Subjects)
Number analyzed (Participants) | 32 | 30 | 31
percentage of subjects | 15.6 [3.0 to 28.2] | 40.0 [22.5 to 57.5] | 32.3 [15.8 to 48.7]

6. Secondary Outcome: Percentage of Subjects Who Achieve CDAI Response at Week 4
Description: CDAI Response at Week 4 is defined as clinical response at Week 4 or remission at Week 4. Clinical response is defined as at least a 100-point decrease from the Week 0 CDAI score, where change = (CDAI score at Week 4) - (CDAI score at Week 0). Remission is defined as a CDAI score of <= 150 points.
Time Frame: Baseline, Week 4
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Full Analysis Set (Placebo Treated Subjects) | Full Analysis Set (CZP 200 mg Treated Subjects) | Full Analysis Set (CZP 400 mg Treated Subjects)
Number analyzed (Participants) | 32 | 30 | 31
percentage of subjects | 21.9 [7.6 to 36.2] | 46.7 [28.8 to 64.5] | 38.7 [21.6 to 55.9]

7. Secondary Outcome: Percentage of Subjects Who Achieve a Reduction in CDAI Scores of at Least 70 Points at Week 2
Description: The Crohn's Disease Activity Index (CDAI) is used to quantify the symptoms of subjects with Crohn's Disease. A score of 150 or below indicates disease remission and a score above 450 indicates extremely severe disease. A decrease in CDAI over time indicates improvement in disease activity.
Time Frame: Baseline, Week 2
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Full Analysis Set (Placebo Treated Subjects) | Full Analysis Set (CZP 200 mg Treated Subjects) | Full Analysis Set (CZP 400 mg Treated Subjects)
Number analyzed (Participants) | 32 | 30 | 31
percentage of subjects | 28.1 [12.5 to 43.7] | 46.7 [28.8 to 64.5] | 45.2 [27.6 to 62.7]

8. Secondary Outcome: Percentage of Subjects Who Achieve a Reduction in CDAI Scores of at Least 70 Points at Week 4
Description: as for outcome 7
Time Frame: Baseline, Week 4
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Full Analysis Set (Placebo Treated Subjects) | Full Analysis Set (CZP 200 mg Treated Subjects) | Full Analysis Set (CZP 400 mg Treated Subjects)
Number analyzed (Participants) | 32 | 30 | 31
percentage of subjects | 25.0 [10.0 to 40.0] | 56.7 [38.9 to 74.4] | 54.8 [37.3 to 72.4]

9. Secondary Outcome: Percentage of Subjects Who Achieve a Reduction in CDAI Scores of at Least 70 Points at Week 6
Description: as for outcome 7
Time Frame: Baseline, Week 6
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Full Analysis Set (Placebo Treated Subjects) | Full Analysis Set (CZP 200 mg Treated Subjects) | Full Analysis Set (CZP 400 mg Treated Subjects)
Number analyzed (Participants) | 32 | 30 | 31
percentage of subjects | 43.8 [26.6 to 60.9] | 53.3 [35.5 to 71.2] | 61.3 [44.1 to 78.4]

10. Secondary Outcome: Percentage of Subjects Who Achieve Remission (CDAI <= 150) at Week 2
Description: Remission at Week 2 is defined as a CDAI score <= 150 points at Week 2.
Time Frame: Week 2
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Full Analysis Set (Placebo Treated Subjects) | Full Analysis Set (CZP 200 mg Treated Subjects) | Full Analysis Set (CZP 400 mg Treated Subjects)
Number analyzed (Participants) | 32 | 30 | 31
percentage of subjects | 3.1 [0.0 to 9.2] | 20.0 [5.7 to 34.3] | 16.1 [3.2 to 29.1]

11. Secondary Outcome: Percentage of Subjects Who Achieve Remission (CDAI <= 150) at Week 4
Description: Remission at Week 4 is defined as a CDAI score <= 150 points at Week 4.
Time Frame: Week 4
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Full Analysis Set (Placebo Treated Subjects) | Full Analysis Set (CZP 200 mg Treated Subjects) | Full Analysis Set (CZP 400 mg Treated Subjects)
Number analyzed (Participants) | 32 | 30 | 31
percentage of subjects | 6.3 [0.0 to 14.6] | 26.7 [10.8 to 42.5] | 22.6 [7.9 to 37.3]

12. Secondary Outcome: Percentage of Subjects Who Achieve Remission (CDAI <= 150) at Week 6
Description: Remission at Week 6 is defined as a CDAI score <= 150 points at Week 6.
Time Frame: Week 6
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Full Analysis Set (Placebo Treated Subjects) | Full Analysis Set (CZP 200 mg Treated Subjects) | Full Analysis Set (CZP 400 mg Treated Subjects)
Number analyzed (Participants) | 32 | 30 | 31
percentage of subjects | 15.6 [3.0 to 28.2] | 26.7 [10.8 to 42.5] | 32.3 [15.8 to 48.7]

13. Secondary Outcome: Percentage of Subjects Who Achieve Clinical Response (Reduction in CDAI Scores of at Least 100 Points) at Week 2
Description: Clinical response is defined as at least a 100-point decrease from the Week 0 CDAI score, where change = (CDAI score at Week 2) - (CDAI score at Week 0).
Time Frame: Baseline, Week 2
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Full Analysis Set (Placebo Treated Subjects) | Full Analysis Set (CZP 200 mg Treated Subjects) | Full Analysis Set (CZP 400 mg Treated Subjects)
Number analyzed (Participants) | 32 | 30 | 31
percentage of subjects | 15.6 [3.0 to 28.2] | 36.7 [19.4 to 53.9] | 29.0 [13.1 to 45.0]

14. Secondary Outcome: Percentage of Subjects Who Achieve Clinical Response (Reduction in CDAI Scores of at Least 100 Points) at Week 4
Description: Clinical response is defined as at least a 100-point decrease from the Week 0 CDAI score, where change = (CDAI score at Week 4) - (CDAI score at Week 0).
Time Frame: Baseline, Week 4
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Full Analysis Set (Placebo Treated Subjects) | Full Analysis Set (CZP 200 mg Treated Subjects) | Full Analysis Set (CZP 400 mg Treated Subjects)
Number analyzed (Participants) | 32 | 30 | 31
percentage of subjects | 18.8 [5.2 to 32.3] | 36.7 [19.4 to 53.9] | 32.3 [15.8 to 48.7]

15. Secondary Outcome: Percentage of Subjects Who Achieve Clinical Response (Reduction in CDAI Scores of at Least 100 Points) at Week 6
Description: Clinical response is defined as at least a 100-point decrease from the Week 0 CDAI score, where change = (CDAI score at Week 6) - (CDAI score at Week 0).
Time Frame: Baseline, Week 6
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Full Analysis Set (Placebo Treated Subjects) | Full Analysis Set (CZP 200 mg Treated Subjects) | Full Analysis Set (CZP 400 mg Treated Subjects)
Number analyzed (Participants) | 32 | 30 | 31
percentage of subjects | 21.9 [7.6 to 36.2] | 36.7 [19.4 to 53.9] | 41.9 [24.6 to 59.3]

16. Secondary Outcome: Inflammatory Bowel Disease Questionnaire (IBDQ) Global Score at Week 2
Description: The IBDQ global score is calculated as the sum of the responses (each ranging from 1 to 7) to all 32 questions on the IBDQ and can therefore range from 32 to 224. A higher score indicates a better quality of life.
Time Frame: Week 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Full Analysis Set (Placebo Treated Subjects) | Full Analysis Set (CZP 200 mg Treated Subjects) | Full Analysis Set (CZP 400 mg Treated Subjects)
Number analyzed (Participants) | 29 | 29 | 31
units on a scale | 171.3 (22.45) | 166.1 (22.14) | 169.7 (23.24)

17. Secondary Outcome: Inflammatory Bowel Disease Questionnaire (IBDQ) Global Score at Week 4
Description: as for outcome 16
Time Frame: Week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Full Analysis Set (Placebo Treated Subjects) | Full Analysis Set (CZP 200 mg Treated Subjects) | Full Analysis Set (CZP 400 mg Treated Subjects)
Number analyzed (Participants) | 28 | 27 | 30
units on a scale | 172.6 (24.04) | 169.4 (21.75) | 170.3 (23.72)

18. Secondary Outcome: Inflammatory Bowel Disease Questionnaire (IBDQ) Global Score at Week 6
Description: as for outcome 16
Time Frame: Week 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Full Analysis Set (Placebo Treated Subjects) | Full Analysis Set (CZP 200 mg Treated Subjects) | Full Analysis Set (CZP 400 mg Treated Subjects)
Number analyzed (Participants) | 28 | 27 | 30
units on a scale | 173.1 (25.49) | 165.6 (23.25) | 170.8 (24.54)

19. Secondary Outcome: Inflammatory Bowel Disease Questionnaire (IBDQ) Domain Scores at Week 2
Description: The total IBDQ score consists of 32 questions, each ranging from 1 to 7, with higher scores indicating a better quality of life.
  There are 4 IBDQ Domain Scores:
  * Bowel Symptoms Domain Score, ranging from 10 to 70 (10 questions ranging from 1 to 7)
  * Systemic Symptoms Domain Score, ranging from 5 to 35 (5 questions ranging from 1 to 7 )
  * Emotional Function Domain Score, ranging from 12 to 84 (12 questions ranging from 1 to 7)
  * Social Function Domain Score, ranging from 5 to 35 (5 questions ranging from 1 to 7 )
Time Frame: Week 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Full Analysis Set (Placebo Treated Subjects) | Full Analysis Set (CZP 200 mg Treated Subjects) | Full Analysis Set (CZP 400 mg Treated Subjects)
Number analyzed (Participants) | 32 | 30 | 31
units on a scale
  Bowel Symptoms Domain Score: number analyzed (Participants) | 29 | 29 | 31
  Bowel Symptoms Domain Score | 54.4 (7.17) | 53.4 (8.18) | 54.7 (8.77)
  Systemic Symptoms Domain Score: number analyzed (Participants) | 29 | 29 | 31
  Systemic Symptoms Domain Score | 22.4 (5.01) | 22.4 (5.17) | 22.7 (4.51)
  Emotional Function Domain Score: number analyzed (Participants) | 29 | 29 | 31
  Emotional Function Domain Score | 65.3 (8.91) | 62.3 (9.54) | 63.3 (8.53)
  Social Function Domain Score: number analyzed (Participants) | 28 | 29 | 31
  Social Function Domain Score | 29.4 (5.64) | 28.0 (4.33) | 29.0 (5.03)

20. Secondary Outcome: Inflammatory Bowel Disease Questionnaire (IBDQ) Domain Scores at Week 4
Description: as for outcome 19
Time Frame: Week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Full Analysis Set (Placebo Treated Subjects) | Full Analysis Set (CZP 200 mg Treated Subjects) | Full Analysis Set (CZP 400 mg Treated Subjects)
Number analyzed (Participants) | 32 | 30 | 31
units on a scale
  Bowel Symptoms Domain Score: number analyzed (Participants) | 28 | 27 | 30
  Bowel Symptoms Domain Score | 55.4 (7.22) | 54.0 (9.00) | 55.5 (8.04)
  Systemic Symptoms Domain Score: number analyzed (Participants) | 28 | 27 | 30
  Systemic Symptoms Domain Score | 23.3 (5.49) | 23.4 (4.21) | 22.9 (4.44)
  Emotional Function Domain Score: number analyzed (Participants) | 28 | 27 | 30
  Emotional Function Domain Score | 65.3 (8.85) | 63.1 (8.90) | 63.2 (9.55)
  Social Function Domain Score: number analyzed (Participants) | 27 | 27 | 30
  Social Function Domain Score | 28.8 (6.73) | 28.9 (4.82) | 28.7 (5.62)

21. Secondary Outcome: Inflammatory Bowel Disease Questionnaire (IBDQ) Domain Scores at Week 6
Description: as for outcome 19
Time Frame: Week 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Full Analysis Set (Placebo Treated Subjects) | Full Analysis Set (CZP 200 mg Treated Subjects) | Full Analysis Set (CZP 400 mg Treated Subjects)
Number analyzed (Participants) | 32 | 30 | 31
units on a scale
  Bowel Symptoms Domain Score: number analyzed (Participants) | 28 | 27 | 30
  Bowel Symptoms Domain Score | 55.4 (7.77) | 51.8 (8.44) | 55.8 (8.43)
  Systemic Symptoms Domain Score: number analyzed (Participants) | 28 | 27 | 30
  Systemic Symptoms Domain Score | 23.3 (6.74) | 22.4 (4.49) | 23.4 (4.62)
  Emotional Function Domain Score: number analyzed (Participants) | 28 | 27 | 30
  Emotional Function Domain Score | 65.3 (8.76) | 63.2 (9.45) | 62.1 (10.43)
  Social Function Domain Score: number analyzed (Participants) | 27 | 27 | 30
  Social Function Domain Score | 29.2 (6.48) | 28.1 (5.69) | 29.5 (5.09)

22. Secondary Outcome: Concentration of C-reactive Protein (CRP) Value at Week 2
Description: CRP data for subjects receiving rescue medication were excluded.
Time Frame: Week 2
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mg/L
Arm/Group | Full Analysis Set (Placebo Treated Subjects) | Full Analysis Set (CZP 200 mg Treated Subjects) | Full Analysis Set (CZP 400 mg Treated Subjects)
Number analyzed (Participants) | 29 | 29 | 31
mg/L | 22.15 [15.43 to 31.80] | 13.58 [9.45 to 19.52] | 13.86 [9.11 to 21.09]

23. Secondary Outcome: Concentration of C-reactive Protein (CRP) Value at Week 4
Description: CRP data for subjects receiving rescue medication were excluded.
Time Frame: Week 4
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mg/L
Arm/Group | Full Analysis Set (Placebo Treated Subjects) | Full Analysis Set (CZP 200 mg Treated Subjects) | Full Analysis Set (CZP 400 mg Treated Subjects)
Number analyzed (Participants) | 28 | 27 | 30
mg/L | 23.47 [16.02 to 34.40] | 12.87 [8.56 to 19.36] | 12.02 [8.68 to 16.65]

24. Secondary Outcome: Concentration of C-reactive Protein (CRP) Value at Week 6
Description: CRP data for subjects receiving rescue medication were excluded.
Time Frame: Week 6
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mg/L
Arm/Group | Full Analysis Set (Placebo Treated Subjects) | Full Analysis Set (CZP 200 mg Treated Subjects) | Full Analysis Set (CZP 400 mg Treated Subjects)
Number analyzed (Participants) | 28 | 27 | 30
mg/L | 23.32 [16.95 to 32.07] | 15.10 [9.46 to 24.11] | 12.62 [8.79 to 18.11]

25. Secondary Outcome: C-reactive Protein (CRP) Ratio to Baseline at Week 2
Description: CRP data for subjects receiving rescue medication were excluded.
Time Frame: Baseline, Week 2
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Full Analysis Set (Placebo Treated Subjects) | Full Analysis Set (CZP 200 mg Treated Subjects) | Full Analysis Set (CZP 400 mg Treated Subjects)
Number analyzed (Participants) | 29 | 29 | 31
ratio | 0.85 [0.64 to 1.13] | 0.58 [0.42 to 0.80] | 0.50 [0.35 to 0.72]

26. Secondary Outcome: C-reactive Protein (CRP) Ratio to Baseline at Week 4
Description: CRP data for subjects receiving rescue medication were excluded.
Time Frame: Baseline, Week 4
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Full Analysis Set (Placebo Treated Subjects) | Full Analysis Set (CZP 200 mg Treated Subjects) | Full Analysis Set (CZP 400 mg Treated Subjects)
Number analyzed (Participants) | 28 | 27 | 30
ratio | 1.04 [0.83 to 1.31] | 0.53 [0.37 to 0.76] | 0.44 [0.32 to 0.60]

27. Secondary Outcome: C-reactive Protein (CRP) Ratio to Baseline at Week 6
Description: CRP data for subjects receiving rescue medication were excluded.
Time Frame: Baseline, Week 6
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Full Analysis Set (Placebo Treated Subjects) | Full Analysis Set (CZP 200 mg Treated Subjects) | Full Analysis Set (CZP 400 mg Treated Subjects)
Number analyzed (Participants) | 28 | 27 | 30
ratio | 1.03 [0.85 to 1.25] | 0.63 [0.40 to 0.98] | 0.46 [0.32 to 0.66]

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from the time of signing the informed consent through the last Observation (up to 28 weeks).
Description: Adverse Events refer to the Safety Population, including all randomized subjects who received at least one dose of study medication (Placebo or Certolizumab Pegol).
Arm/Group | Placebo | Certolizumab Pegol 200 mg | Certolizumab Pegol 400 mg
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/30 | 0/32
Serious Adverse Events (participants affected / at risk) | 3/32 | 1/30 | 3/32
Other Adverse Events (participants affected / at risk) | 16/32 | 11/30 | 14/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=32) | Certolizumab Pegol 200 mg (N=30) | Certolizumab Pegol 400 mg (N=32)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Crohn's disease (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Peritonitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 2 (2)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=32) | Certolizumab Pegol 200 mg (N=30) | Certolizumab Pegol 400 mg (N=32)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (3) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (3) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 2 (3) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 10 (11) | 7 (8) | 7 (9)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1)
Pharynx discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2)
Comedone (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days